CLINICAL TRIAL: NCT04317352
Title: Distal Pancreatectomy With Multivisceral Resection: A Multicentric Study
Brief Title: Multivisceral Resection in Distal Pancreatectomy
Acronym: ERPANDIS-MRV
Status: Completed | Type: Observational
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Gerardo Blanco-Fernández, Chief of department, Universidad de Extremadura
Other Study IDs: UE-CHU 003-2020
Record Dates: First submitted 2020-03-19; First posted 2020-03-23 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Pancreatic Neoplasms; Surgical Procedure, Unspecified
Keywords: Complications; distal pancreatectomy; Multivisceral; resection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multivisceral resection (MRV): MVR: Multivisceral resection was considered when the exeresis of an organ other than the pancreatic body-tail and / or spleen was performed.
  Interventions: Procedure: MVR

INTERVENTIONS:
Procedure: MVR — Multivisceral resection was considered when the exeresis of an organ other than the pancreatic body-tail and / or spleen was performed.

SUMMARY:
The objective of the study is to evaluate the characteristics of the patients and the results of morbidity and mortality after distal pancreatectomy isolated or accompanied by multivisceral resection including cholecystectomy.

DETAILED DESCRIPTION:
Multicenter study that includes patients operated on for distal pancreatectomy between January 2009 to December 2019 for primary pancreatic tumors. Both open or laparoscopic approaches are considered in the study. The objective is to evaluate the characteristics of the patients and the results of morbidity and mortality after distal pancreatectomy isolated or accompanied by multivisceral resection including cholecystectomy. For this, demographic data, variables related to the tumor, surgical intervention and postoperative evolution were collected.

Definitions:

Diagnosis was based mainly on computed tomography (CT scan), Magnetic Resonance (MRI) and endoscopic ultrasonography (USE) plus biopsy. Surgical technique includes open and laparoscopic approach with or without spleen preservation. Complications were assessed at 90 days using the Clavien - Dindo classification, and those defined as Clavien - Dindo grade IIIA or higher were considered major. For the recording of complications, the medical and nursing notes of the electronic or histories of each patient were consulted. For the specific complications of pancreatic surgery, the definitions of the International Study Group on Pancreatic Surgery (ISGPS) of delayed gastric emptying (21), post-pancreatic hemorrhage (22) and pancreatic fistula were used. The resection margins of the surgical specimen were categorized according to the definitions of the Royal College of Pathologists: R0 (margin to the tumor ≥ 1mm), R1 (margin to the tumor <1mm) and R2 (macroscopically positive margin) (24). Tumors were staged according to the TNM classification 8 º Ed. (TNM). Follow up scheme was: 6-month outpatient clinic visit during first five years including tumoral markers and CT/MRI. After five years only once a year visit policy was applied.

Variables The following variables were studied: Epidemiological: age, sex, past medical history, medication, Charlson Index and American Society of Anesthesiology (ASA) classification; Clinical: symptoms due to mucinous neoplasm (MCN); Serological tests: leukocytes, amylase; hemoglobin (gr/dl), bilirubin, creatinin, prothrombin time, carcinoembryonic antigen (CEA) and carbohydrate antigen (CA) 19-9; Radiological/diagnostic: diagnostic tests performed (CT/MRI/EUS), number, size and location of MCN, vascular infiltration (arterial and venous) and preoperative biopsy; Surgical: type of approach (open/laparoscopy/conversion), spleen preservation, associated procedures (organs resected), type of closure of pancreatic remnant, intraoperative bleeding (ml); postoperative course: morbidity and mortality (according to the Clavien-Dindo (CD) classification) (13), pancreatic fistula, postoperative hemorrhage and delayed gastric empting, if present, was classified according to the International Group Study Pancreatic Surgery (IGSPS) classification (14,15), hospital stay and readmissions. The histological data retrieved were TNM: tumor size and lymph nodes harvested and R status. Postoperative follow-up (months) including endocrine and exocrine insufficiency rate.

ELIGIBILITY:
Inclusion Criteria:

* Any distal pancreatectomy (DP) with multivisceral resection (MVR) defining MVR as any organ different from distal pancreas or spleen

Exclusion Criteria:

* Distal Pancreatectomy with celiac trunk resection (Appleby procedure) or portal vein resection.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing distal pancreatectomy for primary pancreatic tumor at participating centers during the period from January 2009 to December 2018
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
Morbidity | 90 days
  Any complication in the postoperative period
Mortality | 90 days
  If the patient dies in the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: José Manuel Ramia, MD, PhD, Study Director — Hospital Universitario de Guadalajara
Locations (1):
- Universidad de Extremadura- Facultad de Medicina, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The study data will be available upon request to the principal investigator via e-mail.

REFERENCES:
- [Background] Malinka T, Klein F, Andreou A, Pratschke J, Bahra M. Distal Pancreatectomy Combined with Multivisceral Resection Is Associated with Postoperative Complication Rates and Survival Comparable to Those After Standard Procedures. J Gastrointest Surg. 2018 Sep;22(9):1549-1556. doi: 10.1007/s11605-018-3804-z. Epub 2018 May 10. PMID 29748738
- [Background] Burdelski CM, Reeh M, Bogoevski D, Gebauer F, Tachezy M, Vashist YK, Cataldegirmen G, Yekebas E, Izbicki JR, Bockhorn M. Multivisceral resections in pancreatic cancer: identification of risk factors. World J Surg. 2011 Dec;35(12):2756-63. doi: 10.1007/s00268-011-1263-8. PMID 21938586
- [Background] Panzeri F, Marchegiani G, Malleo G, Malpaga A, Maggino L, Marchese T, Salvia R, Bassi C, Butturini G. Distal pancreatectomy associated with multivisceral resection: results from a single centre experience. Langenbecks Arch Surg. 2017 May;402(3):457-464. doi: 10.1007/s00423-016-1514-0. Epub 2016 Oct 27. PMID 27787606
- [Background] Irani JL, Ashley SW, Brooks DC, Osteen RT, Raut CP, Russell S, Swanson RS, Whang EE, Zinner MJ, Clancy TE. Distal pancreatectomy is not associated with increased perioperative morbidity when performed as part of a multivisceral resection. J Gastrointest Surg. 2008 Dec;12(12):2177-82. doi: 10.1007/s11605-008-0605-9. Epub 2008 Aug 2. PMID 18677539
- [Background] Song KB, Kwon J, Kim YW, Hwang DW, Lee JH, Hong S, Lee JW, Hwang K, Yoo D, Kim SC. Prognostic value of adjacent organ resection in patients with left-sided pancreatic ductal adenocarcinoma following distal pancreatectomy. J Hepatobiliary Pancreat Sci. 2019 Jun;26(6):227-234. doi: 10.1002/jhbp.627. Epub 2019 May 11. PMID 30980486
- [Background] Nikfarjam M, Sehmbey M, Kimchi ET, Gusani NJ, Shereef S, Avella DM, Staveley-O'Carroll KF. Additional organ resection combined with pancreaticoduodenectomy does not increase postoperative morbidity and mortality. J Gastrointest Surg. 2009 May;13(5):915-21. doi: 10.1007/s11605-009-0801-2. Epub 2009 Feb 7. PMID 19198960
- [Derived] Ramia JM, Del Rio-Martin JV, Blanco-Fernandez G, Cantalejo-Diaz M, Rotellar-Sastre F, Sabater-Orti L, Carabias-Hernandez A, Manuel-Vazquez A, Hernandez-Rivera PJ, Jaen-Torrejimeno I, Kalviainen-Mejia HK, Esteban-Gordillo S, Munoz-Forner E, De la Plaza R, Longoria-Dubocq T, De Armas-Conde N, Pardo-Sanchez F, Garces-Albir M, Serradilla-Martin M. Distal pancreatectomy with multivisceral resection: A retrospective multicenter study - Case series. Int J Surg. 2020 Oct;82:123-129. doi: 10.1016/j.ijsu.2020.08.024. Epub 2020 Aug 26. PMID 32860956